CLINICAL TRIAL: NCT03697590
Title: Photodynamic Therapy of Actinic Keratosis of the Face and Scalp With and Without Prior Curettage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida M. Heerfordt, Principal investigator, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDT with and without curettage
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-06

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic | interventions — Curettage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDT with no curettage (Experimental)
  Interventions: Drug: No curettage
- Standard PDT (Active Comparator)
  Interventions: Drug: Curettage

INTERVENTIONS:
Drug: No curettage — Standard PDT without curettage
  Arms: PDT with no curettage
Drug: Curettage — Standard PDT
  Arms: Standard PDT

SUMMARY:
Guidelines for photodynamic therapy (PDT) of actinic keratosis recommend pretreatment with curettage. The impact of curettage on the treatment effect is, however, not known. The present study aimed to evaluate whether daylight-PDT without curettage would reduce treatment effect compared to daylight-PDT with curettage.

ELIGIBILITY:
Inclusion Criteria:

- Multiple actinic keratosis on the forehead or scalp

Exclusion Criteria:

* Known allergy to methyl aminolevulinate
* Porphyria
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Complete lesion response rate | Treatment efficacy was evaluated 3 months after PDT
  Complete lesion response rate, was defined as the number of completely responding lesions divided by the total number of treated lesion in each field. Complete lesion response was defined as complete disappearance of the lesion both by palpation and visually.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided